CLINICAL TRIAL: NCT05429541
Title: Pneumococcal Carriage and Serotype Distribution in Children With Otitis Media in Malaysia.
Acronym: OM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IMU University, Malaysia (Other)
Collaborators: International Islamic University Malaysia (Other); Universiti Putra Malaysia (Other); University of Southampton (Other); Merck Sharp & Dohme LLC (Industry); Hospital Serdang (Unknown)
Responsible Party: Principal Investigator, Lokman Hakim Sulaiman, MD, Deputy Vice Chancellor, Research, IMU University, Malaysia
Other Study IDs: MISP #61353
Record Dates: First submitted 2022-06-19; First posted 2022-06-23 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Streptococcus Pneumonia; Otitis Media
MeSH Terms: conditions — Pneumonia; Otitis Media

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Middle ear fluid (MEF) sample and nasopharyngeal swab for cases aged 5 years and below will be cultured and Streptococcus Pneumoniae (Spn) isolates will be inoculated for DNA extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Otitis Media (OM) Case Group: Case definition:
  1. Acute otitis media (AOM)
     AOM will be diagnosed by pneumatic otoscopy by validated otoscopists, when children with acute onset of otalgia had tympanic membranes (TMs) that were:
     1. bulging or full; and
     2. a cloudy or purulent effusion was observed, or the TM was completely opacified; and
     3. TM mobility was reduced or absent
  2. Otitis media with effusion (OME)
     Collection of fluid within the middle ear without signs of acute inflammation, fever or otorrhea. Otoscopic findings include:
     1. dull tympanic membrane (TM)
     2. retraction of TM
     3. fluid level or air bubble
     4. TM colour change
     5. restricted TM mobility with pneumatic otoscopy
  3. Chronic suppurative otitis media (CSOM)
  Otoscopic findings:
  1. Perforated TM
  2. Mucopurulent discharge

SUMMARY:
The purpose of this research is to conduct a multi-center prospective surveillance study focusing upon pneumococcal carriage and serotype epidemiology in patients with otitis media (OM).The data generated will be crucial especially as baseline data for future assessments on the long-term impacts of pneumococcal conjugate vaccine 10 (PCV10) coverage, compared to that of pneumococcal conjugate vaccine 13 (PCV13) that is being used in the majority of other countries. Pneumococcal carriage in patients with OM and serotype distribution will be assessed, including changes in antibiotic resistance. With the establishment of sentinel surveillance in the country, we hope to provide detailed data on the epidemiology of OM in Malaysia; working towards the development of a national surveillance programme for the monitoring of OM burden in the country.

DETAILED DESCRIPTION:
Otitis media (OM) is a condition defined as an inflammation of the middle ear and is one of the most commonly diagnosed infections in children, especially amongst those aged below 5 years (1). By 3 years of age, approximately 80% of children have experienced at least one episode of acute otitis media (AOM) in developed countries. More than 700 million AOM cases are reported annually worldwide at an incidence rate of 10.8%, with Southeast Asia reporting a yearly incidence of 8.2% and disease burden varying substantially by geographical location (2). In Malaysia, based on data published from a population based survey (n=7,041) conducted by the Ministry of Health in 2005 (3),OM with effusion (OME) prevalence was found to be 2.9% amongst individuals all ages, of which 46.5% suffered from hearing loss. Amongst children, OME prevalence was 3.8% in those aged ≤17 years, 1.4% in 13-17 year olds and 2.3% in children ≤12 years of age. The survey also found that prevalence was higher in rural settings (3.2%) compared to urban settings (2.7%). These findings were in contrast to an earlier cross-sectional study based on 5 to 6 years olds from kindergartens in 1993 (n=1,097), where prevalence was 17.9% in the urban district of Kuala Lumpur compared to 9.5% in rural Kuala Selangor (4). AOM was found in Malaysia to have a negative impact on both parental and child quality of life (QoL), with significant indirect healthcare costs and thus substantial economic burden in the population (5).

Studies on the epidemiology of AOM, especially those reliant upon clinical diagnosis and following the uptake of pneumococcal conjugate vaccination (PCV) are few and far between. In Malaysia the prevalence of OME, as described above, has been reported although limited to specific settings and locations, with even fewer assessments on AOM prevalence. Immunisation programmes against Spn have an impact on carriage, and consequently the causative pathogen and infecting strains of Spn in OM infections. There has been a consistent observed association between PCV introduction and a decline of AOM infections caused by Spn. As Malaysia is one of the more recent countries to start the PCV National Immunisation Programme (NIP), this presents an excellent opportunity to begin surveillance on pneumococcal carriage and serotype distribution allowing for a detailed assessment of the epidemiology of OM in the country.

Specific Objectives

1. To determine the prevalence of Streptococcus pneumoniae (Spn) nasopharyngeal carriage among children 5 years of age and below with OM
2. To determine Spn serotypes in children diagnosed with OM

ELIGIBILITY:
Inclusion Criteria:

Children aged ≥3 months and <5 years with clinically diagnosed AOM/CSOM whose parent/legal authorized representative (LAR) is willing to give consent on his/her behalf and attending general practitioner clinics, the ear, nose and throat (ENT) outpatient's department or admitted as a hospital inpatient at hospital sites.

Exclusion Criteria:

Any child aged ≥3 months and <5 years old

* who does not meet the case definition
* whose parent/guardian does not give consent on his/her behalf.
* who had nasal surgery,
* who has chronic respiratory diseases (including asthma) and cardiac condition
* with tympanostomy tubes

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children meeting the inclusion criteria, attending general practitioner clinics, the outpatient department or admitted as hospital inpatients in sentinel teaching hospital sites (International Islamic University Malaysia, Universiti Putra Malaysia and Hospital Serdang). Male and female patients from the three major ethnic groups (Malay, Chinese, and Indian) will be recruited from each sentinel site.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-04-05 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Streptococcus pneumoniae (Spn) nasopharyngeal (NP) carriage among young children with OM (AOM/OME/CSOM). | 12 months
  The absence/presence of nasopharyngeal pneumococcal carriage will be tested using standard bacteriological methods and Streptococcus Pneumoniae (SPN) isolates will be inoculated for DNA extraction and tested by polymerase chain reaction (PCR) for pneumococcal carriage detection.

SECONDARY OUTCOMES:
Serotype distribution of Streptococcus pneumoniae (Spn) among young children with OM (AOM/OME/CSOM). | 12 months
  Spn isolates will be sequenced using whole-genome sequencing (WGS) platform (Illumina, UK) to determine the infecting serotype(s) among children with OM. Serotype and sequence type will be derived from the genomic data using a pipeline to identify the serotype from Illumina WGS reads for given references and multilocus sequence type respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Lokman Hakim Sulaiman, PhD, Principal Investigator — IMU University, Malaysia
Locations (2):
- Malaysia (2):
  - Sultan Ahmad Shah Medical Centre @International Islamic University Malaysia, Kuantan, Pahang
  - Universiti Putra Malaysia, Serdang, Seri Kembangan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mahadevan M, Navarro-Locsin G, Tan HK, Yamanaka N, Sonsuwan N, Wang PC, Dung NT, Restuti RD, Hashim SS, Vijayasekaran S. A review of the burden of disease due to otitis media in the Asia-Pacific. Int J Pediatr Otorhinolaryngol. 2012 May;76(5):623-35. doi: 10.1016/j.ijporl.2012.02.031. Epub 2012 Mar 8. PMID 22404948
- [Background] Monasta L, Ronfani L, Marchetti F, Montico M, Vecchi Brumatti L, Bavcar A, Grasso D, Barbiero C, Tamburlini G. Burden of disease caused by otitis media: systematic review and global estimates. PLoS One. 2012;7(4):e36226. doi: 10.1371/journal.pone.0036226. Epub 2012 Apr 30. PMID 22558393
- [Background] Institute For Public Health. Findings of the National Hearing and Ear Disorders Survey. Malaysia: Institute For Public Health, National Instiutes of Health, Ministry of Health Malaysia; 2009.
- [Background] Saim A, Saim L, Saim S, Ruszymah BH, Sani A. Prevalence of otitis media with effusion amongst pre-school children in Malaysia. Int J Pediatr Otorhinolaryngol. 1997 Jul 18;41(1):21-8. doi: 10.1016/s0165-5876(97)00049-9. PMID 9279632
- [Background] Crawford B, Hashim SS, Prepageran N, See GB, Meier G, Wada K, Coon C, Delgleize E, DeRosa M. Impact of Pediatric Acute Otitis Media on Child and Parental Quality of Life and Associated Productivity Loss in Malaysia: A Prospective Observational Study. Drugs Real World Outcomes. 2017 Mar;4(1):21-31. doi: 10.1007/s40801-016-0099-9. PMID 27888477